CLINICAL TRIAL: NCT00893698
Title: Bilateral Allotransplantation of Upper Limbs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008/17; 2008-A00516-49
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Patients Private of Their Upper Limbs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: bilateral allotransplantation — bilateral allotransplantation of upper limbs

SUMMARY:
The aim of the study is to realize a bilateral transplantation of upper limbs. The first objective is functional but there are aesthetic and psychologic imperatives too. This open and descriptive study needs compatible donor and recipient. The sample should be realized simultaneously and the transplantation should be made by two coordinated teams according to this sequence : osteosynthesis, vascular anastomosis, sutures of tendons and nervous sutures. An immunosuppressant treatment should be initialized from the beginning of the intervention and continued for life. Rejections should be screened by regular clinical and histological examinations.

ELIGIBILITY:
Inclusion Criteria:

Donor:

* State of brain death
* Compatibility with recipient about sex, size, age and color
* Blood compatibility; integrity of upper limbs

Recipient:

* Double amputation of hands or forearms with traumatic origin
* Personal motivation
* Good health condition
* Delay from 2 months to 34 years between amputation and transplantation

Exclusion Criteria:

Donor:

* Uncompatibility with sample
* Lesion on upper limbs
* Neoplasia
* Hepatitis B or C
* Positive CMV serology

Recipient:

* Uncompatibility with immunosuppressant treatment
* Psychosis
* Carcinosis
* Cardiovascular diseases
* Addiction to alcohol or smoking
* Pregnancy
* Feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Functional rehabilitation of patients by bilateral allotransplantation of upper limbs, evaluated by measure of the function of the transplanted extremities | 6 years

SECONDARY OUTCOMES:
Aesthetic and psychologic | 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France